CLINICAL TRIAL: NCT04732715
Title: The CaRE Course: Caregiving and Racial Considerations During a Pandemic Online Training Education
Brief Title: Caregiving and Racial Considerations During a Pandemic Online Training Education
Acronym: CaRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Retirement Research Foundation (Other)
Responsible Party: Principal Investigator, Fayron Epps, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00002078
Record Dates: First submitted 2021-01-27; First posted 2021-02-01 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Caregiver Stress Syndrome
Keywords: Disparities; Black American Caregivers; Dementia Caregiving

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CaRE Course (Experimental): Black American caregivers of PLWD will participate in the CaRE Course.
  Interventions: Behavioral: CaRE Course

INTERVENTIONS:
Behavioral: CaRE Course — Participants will complete the CaRE Course over a 6-8 week time period. The curriculum of the CaRE course will include topics addressing caregiving for a PLWD during a pandemic, navigating the healthcare system for a PLWD, guiding and managing daily life, and self care.

SUMMARY:
The overall goal of this project is to develop and prototype-test a highly accessible program designed to enhance the mastery of Black American caregivers to provide care to family members or friends living with a dementia illness in a time of crisis. Participants will be asked a series of questions in a baseline interview, and then will be asked to partake in the CaRE course during a 6 to 8-week period.

DETAILED DESCRIPTION:
Black Americans have over double the prevalence of Alzheimer's disease and related dementias (ADRD) compared to Whites, thus increasing the number of family members providing care for a person living with dementia (PLWD) within this racial/ethnic group. Black American caregivers typically deal with the complexities of caregiving through the lens of race and associated health disparities. Due to the centuries-old disadvantaged social history of Black Americans, a number of unique stressors, vulnerabilities, but also resources, have emerged which could inform and affect Black American dementia caregivers' experiences and well-being. There is overwhelming evidence that Black American caregivers and their care recipients experience disparities in care, have lower rates of formal service use, and are generally under-treated. Now in this seemingly worst of times with the coronavirus disease 2019 (COVID-19) pandemic, the disparities are more apparent: Black Americans (13.4% of the population according to the 2019 U.S. Census Bureau), account for approximately 25% of COVID-19 related deaths and are dying at a rate more than 1.5 times higher than their counterparts. The proposed CaRE Course is meant to address the cultural reality of caregiving while Black - not just during the pandemic, but beyond. The program seeks to develop caregiving mastery while and by understanding, acknowledging, and addressing the influence of race, culture, and disparities on caregivers' mental health, and their medical, spiritual, and safety needs.

The researchers will first establish a preliminary competency-based course curriculum storyboard of 40-50 modules and draft scripts for the instructional videos that will anchor the CaRE course, through iterative Design Studio sessions with Black faith and community leaders, Black American caregivers, course faculty, COVID-19 specialists, dementia experts, and other clinical experts and working with Emory Nursing Experience instructional designers. Then, partnering with a variety of faith-based and community organizations and others, the researchers will identify a sample of Black American caregivers who will be invited to enroll in the CaRE Course and participate in formative and summative research related to its usability, salience, and preliminary efficacy.

ELIGIBILITY:
Inclusion Criteria:

* self-identify as Black American
* unpaid principal caregiver of a community-dwelling person living with a dementing illness and who is the principal companion of that person during healthcare encounters
* provide at least some hands-on care multiple times a week, if not daily
* access to and ability to use broadband internet services to engage with the CaRE Course
* not planning to move the person living with the dementing illness to an institutional setting within the next six months

Exclusion Criteria:

* cannot provide consent
* prisoners
* cognitively impaired adults
* not able to clearly understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Change in Cultural Justification for Caregiving Scale Score | Baseline, Week 10, Week 18
  The Cultural Justification for Caregiving Scale is a 10-item self-report assessing the cultural reasons for the caregivers providing care. Responses are given on a 4-point scale where 1 = strongly disagree and 4 = strongly agree. Total scores range from 10 to 40 with higher scores indicating greater cultural influences for providing care.
Change in Center for Epidemiologic Studies (CES)-Depression Scale Score | Baseline, Week 10, Week 18
  The CES - Depression scale is a 20-item self-report instrument assessing how often symptoms of depression have been experienced in the last week. For this study, responses are given on a 4-point scale where 1 = rarely or none of the time and 4 = most or all of the time. Total scores range from 20 to 80 where higher scores indicate greater caregiver depression.
Change in State-Trait Anxiety Inventory (STAI) Y Form Score | Baseline, Week 10, Week 18
  The STAI Y Form is a 20-item self-report scale of positive and negative anxiety experiences. Responses are given on a 4-point scale where 1 = not at all and 4 = very much so. Total scores range from 20 to 80 where higher scores indicate greater anxiety.
Change in Perceived Stress Scale Score | Baseline, Week 10, Week 18
  The Perceived Stress Scale is a14-item scale assessing the caregivers' feelings and thoughts during the past month. Responses are given on a 5-point scale where 0 = never and 4 = very often. Total scores range from 0 to 40 where higher scores indicate greater perceived stress.
Change in Revised Memory and Behavior Problem Checklist (RMBPC) Score | Baseline, Week 10, Week 18
  The RMBPC is a 24-item scale assessing the frequency of problems that persons with dementia often have as well as how much these behaviors bothered the caregiver. Caregiver reactions are assessed on a 5-point scale where 0 = not at all upset and 4 = extremely upset. Total scores range from 0 to 96 where higher scores indicate greater caregiver distress in reaction to problem behaviors.
Change in Zarit Burden Interview Score | Baseline, Week 10, Week 18
  The Zarit Burden Interview is a 22-item instrument assessing objective and subjective caregiver burden. Responses are given on a 5-point scale where 0 = never and 4 = nearly always. Total scores range from 0 to 88 where higher scores indicate greater feelings of being burdened by being a caregiver.
Change in Caregiver Mastery Score | Baseline, Week 10, Week 18
  The Caregiver Mastery instrument includes 14-items assessing feelings experienced as a result of being a caregiver to a person with dementia. The instrument includes categories of relational deprivation, caregiving competence, and management of situations. Responses are given on a 4-point scale where 1 = not at all and 4 = completely. Total scores range from 14 to 56, where higher scores indicate feeling a greater sense of mastery of caregiving.

CONTACTS AND LOCATIONS:
Overall Officials: Fayron Epps, PhD, RN, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial will be made available for sharing, after deidentification.
Supporting Information: Study Protocol
Time Frame: Data will be made available for sharing beginning 3 months and ending 5 years following article publication.
Access Criteria: Data will be made available for sharing with researchers who provide a methodologically sound proposal, in order to achieve aims in the approved proposal. Proposals should be directed to fepps@emory.edu. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years via a third party website.